CLINICAL TRIAL: NCT06953648
Title: Remotely Monitored, Mobile Health-supported, High Intensity Interval Training Before Hematopoietic Stem Cell Transplantation (REMM-HIIT-HCT)
Brief Title: Remotely Monitored, Mobile Health-supported, High Intensity Interval Training Before Hematopoietic Stem Cell Transplant
Acronym: REMM-HIIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REMM-HIIT
Record Dates: First submitted 2025-03-26; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Stem Cell Transplantation; Cardiorespiratory Fitness
Keywords: High Intensity Interval Training; HIIT; Hematopoietic Stem Cell Transplantation; Remote Monitoring; Mobile Health; Exercise; Cardiorespiratory Fitness
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Group (Experimental): The intervention will consist of three 30-minute training sessions/week, each starting with a five-minute warm-up, followed by 20 minutes of interval training, and ending with a five-minute cool-down. The interval training will consist of 10 alternating high- and low-intensity intervals, with a 1:1 work-to-rest ratio (one minute of high intensity followed by one minute of low-moderate intensity).
  Interventions: Behavioral: High Intensity Interval Training
- Control Group (No Intervention): Participants will receive a handout and information on exercise.

INTERVENTIONS:
Behavioral: High Intensity Interval Training — The intervention will consist of three 30-minute training sessions/week, each starting with a five-minute warm-up, followed by 20 minutes of interval training, and ending with a five-minute cool-down. The interval training will consist of 10 alternating high- and low-intensity intervals, with a 1:1 work-to-rest ratio (one minute of high intensity followed by one minute of low-moderate intensity). As participants' fitness improves, the interval intensity will increase accordingly.
  Arms: HIIT Group

SUMMARY:
The goal of this clinical trial is to learn how a remotely monitored high-intensity interval training (REMM-HIIT) affects the cardiorespiratory fitness and physical function for patients planning to undergo stem cell transplantation. The main questions it aims to answer are:

Is there a change in the participant's cardiorespiratory fitness level? Is there a change in the participant's physical function?

Researchers will compare the REMM-HIIT program to a control group of participants who do not take part in the training program to see if REMM-HIIT helps improve stem cell transplantation outcomes.

Participants will:

* Complete cardiopulmonary exercise testing (CPET) 4 times during the study
* Do basic tests to measure physical function 6 times during the study
* Answer questions about their life and how they are feeling 6 times during the study
* Wear a device to keep track of step counts and heart rate daily
* Keep a log of every time they exercise throughout the study
* Optionally, provide blood and stool samples 6 times during the study

DETAILED DESCRIPTION:
Each year in the U.S., approximately 8,000 patients undergo allogeneic hematopoietic stem cell transplantation (HCT) as a potentially curative therapy for leukemias, lymphomas, and other hematologic malignancies. However, treatment-related mortality (TRM) is significant, ranging from 10-30%. Moreover, survivors of HCT often face significant physical, psychological, and social challenges post-treatment, leading to a substantial decrease in quality of life (QOL). Outcomes are closely linked to pre-HCT physical activity and function. For example, patients with worse pre-HCT physical function and capacity have markedly lower one-year survival rates (50% vs. 83%). In contrast, every 50-meter increase in pre-HCT six-minute walk distance (6MWD) correlates with a 9% reduction in relative risk for mortality.

Cardiorespiratory fitness (CRF) is a crucial indicator of physical capacity, reflecting the integrated functioning of the heart, lungs, skeletal muscle, adipose tissue, pancreas, liver and adrenal tissues. While CRF naturally declines with age, this decline is notably accelerated by cancer and its treatments, with cancer patients' average CRF levels comparable to individuals 20-30 years older. Importantly, patients with low pre-HCT CRF (VO2peak <16 mL/kg/min) are at much higher risk of TRM (hazard ratio 6.70), even after accounting for other risk factors. This underscores the critical need for interventions to improve CRF prior to HCT to enhance survival and post-treatment quality of life.

It is well established that patients with better pre-HCT physical function tend to have better post-HCT outcomes. The critical question, however, is whether enhancing fitness pre-HCT can improve post-HCT outcomes. Animal studies provide optimism: exercise training in a murine model pre-HCT associated with improved survival, possibly through immune-mediated pathways. Yet, research exploring the impact of pre-HCT exercise on human post-HCT outcomes remains limited. Small studies have linked pre-HCT improvements in physical function with better survival, and preliminary results from a randomized controlled trial suggest that exercise during HCT may reduce mortality. However, a recent large (n=711) randomized Blood and Marrow Transplant Clinical Trials Network study of self-directed exercise and stress management during HCT did not show a significant benefit in outcomes. Study investigators suggested several reasons for this lack of effect, including timing of intervention (peri-HCT rather than pre-HCT), low intensity rather than high intensity exercise, and low engagement in the self-directed program.

To address prior study limitations, the investigators developed the REMM-HIIT program, focusing on pre-HCT intervention, high-intensity interval training (HIIT), and a mobile health (mHealth) platform to support participant engagement. This program, supported by the National Institute of Aging and the Duke Claude D. Pepper Older Americans Independence Center, was piloted in a successful phase 1 study of Remotely Monitored, Mobile health-supported, pre-HCT High Intensity Interval Training (REMM-HIIT). In this feasibility study, participants underwent baseline cardiopulmonary exercise testing (CPET) to ensure cardiac safety and to measure maximal cardiorespiratory fitness (VO2peak). The heart rate (HR) at VO2peak was used to personalize the high and low intensity interval goals. Participants were equipped with an iPhone and Garmin Watch for remote monitoring and exercised three times a week at home, with the first session and subsequent sessions as needed monitored remotely by the coach via videoconference. This approach ensured continuous support and maximized participant engagement while allowing the majority of sessions to occur remotely.

This program was purposely designed based on investigators' prior research and other significant studies in the field, aiming to overcome common barriers to physical activity in cancer populations. To facilitate participation, the investigators enable exercise at home utilizing the participant's preferred activity (e.g., walking, cycling, stairs) and at convenient times. The majority engaged in walking-based intervention, which despite their simplicity, provided sufficient intensity for deconditioned HCT participants. Others used cycle ergometers. This program adheres to the principles of exercise training and recommendations from Sasso and colleagues, ensuring individualization, progressive overload, appropriate recovery periods, and reasonable specificity. Exercise sessions started with a 5-minute warmup (e.g., walking or cycling at a HR corresponding to 60% VO2peak). This was followed by ten intervals, each consisting of one-minute of high intensity exercise at a HR corresponding to 95% VO2peak, alternated with one minute of low to moderate intensity interval at a HR corresponding to 60% VO2peak, totaling 20 minutes. The session concluded with a 5-minute cooldown, resulting in a comprehensive 30-minutes exercise session. For participants unable to complete all intervals, the study team began with fewer intervals and gradually increased the number as tolerated. A recovery period of 24-48 hours between HIIT sessions was recommended to prevent overtraining and ensure adequate recovery. Broad specificity was achieved by incorporating high, moderate, and low intensity aerobic exercises continuously. As such, the program is a progressive HIIT-based intervention, with flexibility given to ensure the principles of exercise training are upheld, and participants receive the best possible information and guidance to rapidly increase CRF and health outcomes pre-HCT.

The investigators' prior phase 1 study was successful. Out of 24 participants approached, 14 enrolled (10 males, 4 females), achieving a recruitment rate of 58%. Of the 14 enrolled, 13 (age 59±12, range 34-76 yrs; 10 White, 3 Black) were medically cleared to proceed with HIIT following a CPET. One participant did not proceed to HIIT and was withdrawn due to cardiac concerns detected on baseline CPET. Importantly, there were no adverse events associated with exercise among the remaining participants. Participants were able to engage in HIIT, even with a baseline CRF as low as 10.6 mL/kg/min; for reference, independent living in healthy adults is generally associated with a CRF >18 in men and >15 in women. Some participants who were habitually exercising were able to complete ten intervals immediately and to maintain intensity over time, while other participants who were less fit required more coaching but were able to rapidly improve fitness to reach program goals. Remarkably, even with low baseline CRF and concomitant chemotherapy (some requiring hospitalization), nine of the 13 participants engaged in the exercise program (69%), and average adherence to the prescribed 3 sessions/week in those nine was excellent at 104 +/- 28%. Mean intervention length was 13.8 +/- 7.5 weeks, with participants staying engaged in the exercise program for approximately three months prior to HCT; this compares very favorably to the 50-70% adherence rates commonly reported in other home-based exercise studies. All 7 participants who had repeat CPET showed improvements in CRF, with average change in VO2peak from 14.6 ± 3.1 mL/kg/min at enrollment to 17.9 ± 3.3 by the start of transplant, or 23% increase (p<0.001). For the other 6, 3 were not evaluated due to the onset of the COVID-19 pandemic, which suspended research operations. Because CRF declines at about 10% per decade, this substantial improvement in CRF equates to a fitness level increase that typically would take over 20 years to achieve, aligning participants' fitness more closely with that of healthy adults34. As highlighted by Wood et al.,16 a pre-HCT VO2peak <16 mL/kg/min is associated with higher post-HCT mortality rate (HR 6.70 (1.29-34.75), p=0.02) and longer hospital stay (median number of hospitalized days before Day 100: 33 vs. 21, p=0.004). Thus, increasing CRF pre-HCT has the potential to improve post-HCT outcomes, suggesting this program could substantially impact participant health and recovery.

The investigators believe this program's success is from a combination of participant motivation and mHealth platform and coaching. Because participants know that they were to undergo HCT within a few months, with a 10-30% chance of death related to the treatment itself, they were highly motived to do anything they could to improve their chances of survival. Furthermore, knowing that an oncology-experienced exercise professional is monitoring their exercise sessions, coupled with personalized and frequent feedback (at least once a week), likely helped improve adherence, with resultant improvements in CRF.

Allogeneic HCT has curative potential for hematologic malignancies but is associated with significant morbidity and TRM, especially in patients with low pre-HCT CRF. Improving CRF through a time-efficient, high-intensity interval training (HIIT) approach, facilitated remotely via mHealth, could improve physical function and clinical outcomes for HCT patients. The investigators hypothesize that patients undergoing REMM-HIIT program will experience improved CRF, physical function, and QOL pre-HCT, leading to better post-HCT outcomes, including improved physical function, reduced TRM, and increased overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Plan to undergo allogeneic hematopoietic stem cell transplant in 4-12 weeks after enrollment on this study.
* Age 18-80 years
* Able to read/write English (as many participant-reported outcome measures lack validated translations in other languages)

Exclusion Criteria:

* Unable or unwilling to follow coaching
* Functional impairment resulting in inability to exercise
* Any absolute contraindications to exercise:

  1. recent (<6 months) acute cardiac event;
  2. unstable angina;
  3. uncontrolled dysrhythmias causing symptoms;
  4. symptomatic aortic stenosis;
  5. uncontrolled symptomatic heart failure;
  6. acute pulmonary embolus;
  7. acute myocarditis or pericarditis;
  8. suspected or known dissecting aneurysm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | At Baseline, Day -10, Day 90, and Day 365
  Change in cardiorespiratory fitness as measured by the difference in peak rate of oxygen consumption (VO2peak) in mL/(kg*min) from baseline to the pre-hematopoietic stem cell transplant (HCT) timepoint; a higher number for VO2 peak indicates greater cardiorespiratory fitness.
Change in Physical Function (Six Minute Walk Test Distance) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The change in physical function as measured by the difference in six minute walk test distance in meters from baseline to the pre-hematopoietic stem cell transplantation (HCT) timepoint; a greater number of meters walked indicates a higher level of physical function.

SECONDARY OUTCOMES:
Effect on Health-related Quality of Life (Physical Activity/Short Physical Performance Battery) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (physical activity) as measured by performance on the Short Physical Performance Battery, which results in a score from 0 to 12 points, with a higher number indicating better physical performance.
Effect on Health-related Quality of Life (Physical Activity/30-Second Sit-to-Stand Test) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related qulaity of life (physical activity) as measured by the 30-second sit-to-stand test, which measures the number of times an individual can stand up from a chair and sit back down within 30 seconds, with a higher number indicating greater fitness.
Effect on Health-related Quality of Life (Physical Activity/Fried Frailty) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (physical activity) as measured by the Fried Frailty assessment, which results in a score from 0 to 5, with a higher number indicating greater frailty.
Effect on Health-related Quality of Life (Physical Activity/Fall Question) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (physical activity) as measured by the Fall Question, a structured questionnaire asking about any history of falls, with a higher number of falls indicating greater fall risk and physical vulnerability.
Effect on Health-related Quality of Life (Physical Activity/Physical Function Questionnaire) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (physical activity) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function questionnaire, which results in a numerical score between 0 and 100, with a higher number indicating better physical function.
Effect on Health-related Quality of Life (Physical Activity/Fatigue Questionnaire) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (physical activity) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue questionnaire, which results in a numerical score between 0 and 100, with a higher number indicating greater symptom burden.
Effect on Health-related Quality of Life (Physical Activity/International Physical Activity Questionnaire) | At Baseline
  Effect on health-related quality of life (physical activity) as measured by the International Physical Activity Questionnaire, which provides 2 results: a categorical rating of low, moderate, or high activity level, and a number of Metabolic Equivalent of Task (MET) minutes per week, with a higher number indicating a greater amount of physical activity.
Effect on Health-related Quality of Life (Cognitive/Montreal Cognitive Assessment) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (cognitive) as measured by the Montreal Cognitive Assessment (MOCA), which results in a numerical score between 0 and 30, with a higher number indicating better cognitive functioning.
Effect on Health-related Quality of Life (Mental Health/Lorig Self-Efficacy) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (mental health) as measured by the Lorig Self-Efficacy for Managing Chronic Disease Scale, which results in a numerical score between 1 and 10, with a higher number indicating higher self-efficacy.
Effect on Health-related Quality of Life (Mental Health/Depression Scale) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (mental health) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression scale, which results in a numerical value between 8 and 40, with a higher number indicating greater severity of depression.
Effect on Health-related Quality of Life (Mental Health/Anxiety scale) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (mental health) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety scale, which results in a numerical value between 7 and 35, with a higher number indicating greater severity of anxiety.
Effect on Health-related Quality of Life (Weight) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (weight) as measured by the change in patient's body weight in kilograms.
Effect on Health-related Quality of Life (Albumin Level) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (albumin level) as measured by the change in patient's albumin level in grams per deciliter; low serum albumin levels can predict higher cancer mortality.
Effect on Health-related Quality of Life (Nutrition) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (nutrition) as measured by the Patient-Generated Subjective Global Assessment (PG-SGA), which gives 2 results: a numerical score between 0 and 16, where a higher score indicates higher nutritional risk, and a categorical score where A = well nourished, B = moderately malnourished, and C = severely malnourished.
Effect on Health-related Quality of Life (Social Support/Emotional Support) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (social support) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support assessment, which results in a numerical score between 8 and 40, with a higher score indicating a greater level of social participation.
Effect on Health-related Quality of Life (Social Support/Social Isolation) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life (social support) as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation assessment, which results in a numerical score between 6 and 30, with a higher score indicating a greater level of social participation.
Effect on Health-related Quality of Life (EuroQoL-5 Dimension-5 Level) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on health-related quality of life as measured by the EuroQoL-5 Dimension-5 Level (EQ-5D-5L), which results in a 5-digit health state, where each digit is between 1 and 5 (e.g. 12345 or 11111). For each digit, a higher number indicates a greater severity of problems.
Effect on Health-related Quality of Life (Return to Work) | At Day 180 and Day 365
  Effect on health-related quality of life as measured by assessing the patient's return to work as an indicator of recovery.
Effect on Clinical Outcomes (Overall Survival) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on clinical outcomes as measured by overall survival.
Effect on Clinical Outcomes (Treatment-related Mortality) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on clinical outcomes as measured by treatment-related mortality.
Effect on Clinical Outcomes (Incidence of Infection) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on clinical outcomes as measured by incidence of infection.
Effect on Clinical Outcomes (Incidence of Graft-versus-host disease) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on clinical outcomes as measured by incidence of graft versus host disease.
Effect on Clinical Outcomes (Time to Relapse) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  Effect on clinical outcomes as measured by time to relapse.
Length of Stay | At day of hospital discharge
  The length of hospital stay measured in days from time of transplant to time of discharge.

OTHER OUTCOMES:
Effect on Muscle Health (Resting Energy Expenditure) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The effect on muscle health as measured by resting energy expenditure.
Effect on Muscle Health (Intramuscular Adipose Tissue) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The effect on muscle health as measured by amount of intramuscular adipose tissue assessed using biopsied muscle tissue.
Effect on Muscle Health (Glycogen Stores) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The effect on muscle health as measured by amount of glycogen stores in muscle assessed using biopsied muscle tissue.
Effect on Muscle Health (Muscle Mitochondrial Metabolism) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The effect on muscle health as measured by muscle mitochondrial metabolism assessed in biopsied muscle tissue.
Effect on Biomarkers (Analysis of Plasma) | At Baseline, Day -10, Day 30, Day 90, Day 180, and Day 365
  The effect on biomarkers as measured by analysis of plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — The University of Kansas Cancer Center
Locations (3):
- United States (3):
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Duke University, Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCulloch CE, Neuhaus JM. Generalized Linear Mixed Models. Encyclopedia of Biostatistics2005
- [Background] David LA, Maurice CF, Carmody RN, Gootenberg DB, Button JE, Wolfe BE, Ling AV, Devlin AS, Varma Y, Fischbach MA, Biddinger SB, Dutton RJ, Turnbaugh PJ. Diet rapidly and reproducibly alters the human gut microbiome. Nature. 2014 Jan 23;505(7484):559-63. doi: 10.1038/nature12820. Epub 2013 Dec 11. PMID 24336217
- [Background] David LA, Weil A, Ryan ET, Calderwood SB, Harris JB, Chowdhury F, Begum Y, Qadri F, LaRocque RC, Turnbaugh PJ. Gut microbial succession follows acute secretory diarrhea in humans. mBio. 2015 May 19;6(3):e00381-15. doi: 10.1128/mBio.00381-15. PMID 25991682
- [Background] Thompson JC, Ren Y, Romero K, Lew M, Bush AT, Messina JA, Jung SH, Siamakpour-Reihani S, Miller J, Jenq RR, Peled JU, van den Brink MRM, Chao NJ, Shrime MG, Sung AD. Financial incentives to increase stool collection rates for microbiome studies in adult bone marrow transplant patients. PLoS One. 2022 May 4;17(5):e0267974. doi: 10.1371/journal.pone.0267974. eCollection 2022. PMID 35507633
- [Background] Team RC. R: A language and environment for statistical computing Vienna, Austria2014.
- [Background] Xie Y. Dynamic Documents with R and knitr. Chapman & Hall/CRC The R Series. Boca Raton, FL: Chapman & Hall/CRC 2013.
- [Background] LIANG K-Y, ZEGER SL. Longitudinal data analysis using generalized linear models. Biometrika. 1986;73(1):13-22. doi: 10.1093/biomet/73.1.13.
- [Background] Jung SH, Ahn C. Sample size estimation for GEE method for comparing slopes in repeated measurements data. Stat Med. 2003 Apr 30;22(8):1305-15. doi: 10.1002/sim.1384. PMID 12687656
- [Background] Gentleman RC, Carey VJ, Bates DM, Bolstad B, Dettling M, Dudoit S, Ellis B, Gautier L, Ge Y, Gentry J, Hornik K, Hothorn T, Huber W, Iacus S, Irizarry R, Leisch F, Li C, Maechler M, Rossini AJ, Sawitzki G, Smith C, Smyth G, Tierney L, Yang JY, Zhang J. Bioconductor: open software development for computational biology and bioinformatics. Genome Biol. 2004;5(10):R80. doi: 10.1186/gb-2004-5-10-r80. Epub 2004 Sep 15. PMID 15461798
- [Background] Huffman KM, Jessee R, Andonian B, Davis BN, Narowski R, Huebner JL, Kraus VB, McCracken J, Gilmore BF, Tune KN, Campbell M, Koves TR, Muoio DM, Hubal MJ, Kraus WE. Molecular alterations in skeletal muscle in rheumatoid arthritis are related to disease activity, physical inactivity, and disability. Arthritis Res Ther. 2017 Jan 23;19(1):12. doi: 10.1186/s13075-016-1215-7. PMID 28114971
- [Background] Huffman KM, Koves TR, Hubal MJ, Abouassi H, Beri N, Bateman LA, Stevens RD, Ilkayeva OR, Hoffman EP, Muoio DM, Kraus WE. Metabolite signatures of exercise training in human skeletal muscle relate to mitochondrial remodelling and cardiometabolic fitness. Diabetologia. 2014 Nov;57(11):2282-95. doi: 10.1007/s00125-014-3343-4. Epub 2014 Aug 5. PMID 25091629
- [Background] Metzger KE, Rucker Y, Callaghan M, Churchill M, Jovanovic BD, Zembower TR, Bolon MK. The burden of mucosal barrier injury laboratory-confirmed bloodstream infection among hematology, oncology, and stem cell transplant patients. Infect Control Hosp Epidemiol. 2015 Feb;36(2):119-24. doi: 10.1017/ice.2014.38. PMID 25632993
- [Background] Dandoy CE, Kim S, Chen M, Ahn KW, Ardura MI, Brown V, Chhabra S, Diaz MA, Dvorak C, Farhadfar N, Flagg A, Ganguly S, Hale GA, Hashmi SK, Hematti P, Martino R, Nishihori T, Nusrat R, Olsson RF, Rotz SJ, Sung AD, Perales MA, Lindemans CA, Komanduri KV, Riches ML. Incidence, Risk Factors, and Outcomes of Patients Who Develop Mucosal Barrier Injury-Laboratory Confirmed Bloodstream Infections in the First 100 Days After Allogeneic Hematopoietic Stem Cell Transplant. JAMA Netw Open. 2020 Jan 3;3(1):e1918668. doi: 10.1001/jamanetworkopen.2019.18668. PMID 31913492
- [Background] Sung AD, Chao NJ. Concise review: acute graft-versus-host disease: immunobiology, prevention, and treatment. Stem Cells Transl Med. 2013 Jan;2(1):25-32. doi: 10.5966/sctm.2012-0115. Epub 2012 Dec 19. PMID 23283494
- [Background] Campbell SC, Wisniewski PJ, Noji M, McGuinness LR, Haggblom MM, Lightfoot SA, Joseph LB, Kerkhof LJ. The Effect of Diet and Exercise on Intestinal Integrity and Microbial Diversity in Mice. PLoS One. 2016 Mar 8;11(3):e0150502. doi: 10.1371/journal.pone.0150502. eCollection 2016. PMID 26954359
- [Background] Bressa C, Bailen-Andrino M, Perez-Santiago J, Gonzalez-Soltero R, Perez M, Montalvo-Lominchar MG, Mate-Munoz JL, Dominguez R, Moreno D, Larrosa M. Differences in gut microbiota profile between women with active lifestyle and sedentary women. PLoS One. 2017 Feb 10;12(2):e0171352. doi: 10.1371/journal.pone.0171352. eCollection 2017. PMID 28187199
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Denou E, Marcinko K, Surette MG, Steinberg GR, Schertzer JD. High-intensity exercise training increases the diversity and metabolic capacity of the mouse distal gut microbiota during diet-induced obesity. Am J Physiol Endocrinol Metab. 2016 Jun 1;310(11):E982-93. doi: 10.1152/ajpendo.00537.2015. Epub 2016 Apr 26. PMID 27117007
- [Background] Evans CC, LePard KJ, Kwak JW, Stancukas MC, Laskowski S, Dougherty J, Moulton L, Glawe A, Wang Y, Leone V, Antonopoulos DA, Smith D, Chang EB, Ciancio MJ. Exercise prevents weight gain and alters the gut microbiota in a mouse model of high fat diet-induced obesity. PLoS One. 2014 Mar 26;9(3):e92193. doi: 10.1371/journal.pone.0092193. eCollection 2014. PMID 24670791
- [Background] Stein-Thoeringer CK, Nichols KB, Lazrak A, Docampo MD, Slingerland AE, Slingerland JB, Clurman AG, Armijo G, Gomes ALC, Shono Y, Staffas A, Burgos da Silva M, Devlin SM, Markey KA, Bajic D, Pinedo R, Tsakmaklis A, Littmann ER, Pastore A, Taur Y, Monette S, Arcila ME, Pickard AJ, Maloy M, Wright RJ, Amoretti LA, Fontana E, Pham D, Jamal MA, Weber D, Sung AD, Hashimoto D, Scheid C, Xavier JB, Messina JA, Romero K, Lew M, Bush A, Bohannon L, Hayasaka K, Hasegawa Y, Vehreschild MJGT, Cross JR, Ponce DM, Perales MA, Giralt SA, Jenq RR, Teshima T, Holler E, Chao NJ, Pamer EG, Peled JU, van den Brink MRM. Lactose drives Enterococcus expansion to promote graft-versus-host disease. Science. 2019 Nov 29;366(6469):1143-1149. doi: 10.1126/science.aax3760. PMID 31780560
- [Background] Guo H, Chou WC, Lai Y, Liang K, Tam JW, Brickey WJ, Chen L, Montgomery ND, Li X, Bohannon LM, Sung AD, Chao NJ, Peled JU, Gomes ALC, van den Brink MRM, French MJ, Macintyre AN, Sempowski GD, Tan X, Sartor RB, Lu K, Ting JPY. Multi-omics analyses of radiation survivors identify radioprotective microbes and metabolites. Science. 2020 Oct 30;370(6516):eaay9097. doi: 10.1126/science.aay9097. PMID 33122357
- [Background] Schluter J, Peled JU, Taylor BP, Markey KA, Smith M, Taur Y, Niehus R, Staffas A, Dai A, Fontana E, Amoretti LA, Wright RJ, Morjaria S, Fenelus M, Pessin MS, Chao NJ, Lew M, Bohannon L, Bush A, Sung AD, Hohl TM, Perales MA, van den Brink MRM, Xavier JB. The gut microbiota is associated with immune cell dynamics in humans. Nature. 2020 Dec;588(7837):303-307. doi: 10.1038/s41586-020-2971-8. Epub 2020 Nov 25. PMID 33239790
- [Background] Khan N, Lindner S, Gomes ALC, Devlin SM, Shah GL, Sung AD, Sauter CS, Landau HJ, Dahi PB, Perales MA, Chung DJ, Lesokhin AM, Dai A, Clurman A, Slingerland JB, Slingerland AE, Brereton DG, Giardina PA, Maloy M, Armijo GK, Rondon-Clavo C, Fontana E, Bohannon L, Ramalingam S, Bush AT, Lew MV, Messina JA, Littmann E, Taur Y, Jenq RR, Chao NJ, Giralt S, Markey KA, Pamer EG, van den Brink MRM, Peled JU. Fecal microbiota diversity disruption and clinical outcomes after auto-HCT: a multicenter observational study. Blood. 2021 Mar 18;137(11):1527-1537. doi: 10.1182/blood.2020006923. PMID 33512409
- [Background] Peled JU, Gomes ALC, Devlin SM, Littmann ER, Taur Y, Sung AD, Weber D, Hashimoto D, Slingerland AE, Slingerland JB, Maloy M, Clurman AG, Stein-Thoeringer CK, Markey KA, Docampo MD, Burgos da Silva M, Khan N, Gessner A, Messina JA, Romero K, Lew MV, Bush A, Bohannon L, Brereton DG, Fontana E, Amoretti LA, Wright RJ, Armijo GK, Shono Y, Sanchez-Escamilla M, Castillo Flores N, Alarcon Tomas A, Lin RJ, Yanez San Segundo L, Shah GL, Cho C, Scordo M, Politikos I, Hayasaka K, Hasegawa Y, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Jenq RR, Teshima T, Chao NJ, Holler E, Xavier JB, Pamer EG, van den Brink MRM. Microbiota as Predictor of Mortality in Allogeneic Hematopoietic-Cell Transplantation. N Engl J Med. 2020 Feb 27;382(9):822-834. doi: 10.1056/NEJMoa1900623. PMID 32101664
- [Background] Franceschi C, Campisi J. Chronic inflammation (inflammaging) and its potential contribution to age-associated diseases. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1:S4-9. doi: 10.1093/gerona/glu057. PMID 24833586
- [Background] Ariffin H, Azanan MS, Abd Ghafar SS, Oh L, Lau KH, Thirunavakarasu T, Sedan A, Ibrahim K, Chan A, Chin TF, Liew FF, Jeyamogan S, Rosli ES, Baharudin R, Yap TY, Skinner R, Lum SH, Hainaut P. Young adult survivors of childhood acute lymphoblastic leukemia show evidence of chronic inflammation and cellular aging. Cancer. 2017 Nov 1;123(21):4207-4214. doi: 10.1002/cncr.30857. Epub 2017 Jun 27. PMID 28654149
- [Background] Parker D, Sloane R, Pieper CF, Hall KS, Kraus VB, Kraus WE, Huebner JL, Ilkayeva OR, Bain JR, Newby LK, Cohen HJ, Morey MC. Age-Related Adverse Inflammatory and Metabolic Changes Begin Early in Adulthood. J Gerontol A Biol Sci Med Sci. 2019 Feb 15;74(3):283-289. doi: 10.1093/gerona/gly121. PMID 29985987
- [Background] Griesenauer B, Paczesny S. The ST2/IL-33 Axis in Immune Cells during Inflammatory Diseases. Front Immunol. 2017 Apr 24;8:475. doi: 10.3389/fimmu.2017.00475. eCollection 2017. PMID 28484466
- [Background] Adom D, Rowan C, Adeniyan T, Yang J, Paczesny S. Biomarkers for Allogeneic HCT Outcomes. Front Immunol. 2020 Apr 21;11:673. doi: 10.3389/fimmu.2020.00673. eCollection 2020. PMID 32373125
- [Background] Harris AC, Ferrara JL, Braun TM, Holler E, Teshima T, Levine JE, Choi SW, Landfried K, Akashi K, Vander Lugt M, Couriel DR, Reddy P, Paczesny S. Plasma biomarkers of lower gastrointestinal and liver acute GVHD. Blood. 2012 Mar 22;119(12):2960-3. doi: 10.1182/blood-2011-10-387357. Epub 2012 Jan 27. PMID 22286196
- [Background] Meng XQ, Chen XH, Sahebally Z, Xu YN, Yin SY, Wu LM, Zheng SS. Cytokines are early diagnostic biomarkers of graft-versus-host disease in liver recipients. Hepatobiliary Pancreat Dis Int. 2017 Feb;16(1):45-51. doi: 10.1016/s1499-3872(16)60157-1. PMID 28119258
- [Background] Kielsen K, Oostenbrink LVE, von Asmuth EGJ, Jansen-Hoogendijk AM, van Ostaijen-Ten Dam MM, Ifversen M, Heilmann C, Schilham MW, van Halteren AGS, Bredius RGM, Lankester AC, Jol-van der Zijde CM, van Tol MJD, Muller K. IL-7 and IL-15 Levels Reflect the Degree of T Cell Depletion during Lymphopenia and Are Associated with an Expansion of Effector Memory T Cells after Pediatric Hematopoietic Stem Cell Transplantation. J Immunol. 2021 Jun 15;206(12):2828-2838. doi: 10.4049/jimmunol.2001077. Epub 2021 Jun 9. PMID 34108260
- [Background] Siamakpour-Reihani S, Cao F, Lyu J, Ren Y, Nixon AB, Xie J, Bush AT, Starr MD, Bain JR, Muehlbauer MJ, Ilkayeva O, Byers Kraus V, Huebner JL, Chao NJ, Sung AD. Evaluating immune response and metabolic related biomarkers pre-allogenic hematopoietic stem cell transplant in acute myeloid leukemia. PLoS One. 2022 Jun 14;17(6):e0268963. doi: 10.1371/journal.pone.0268963. eCollection 2022. PMID 35700185
- [Background] Randall J, Anderson G, Kayser K. Psychosocial assessment of candidates for hematopoietic cell transplantation: A national survey of centers' practices. Psychooncology. 2022 Jul;31(7):1253-1260. doi: 10.1002/pon.5919. Epub 2022 Mar 16. PMID 35278265
- [Background] Stickney Ferguson S, Randall J, Dabney J, Kalbacker ME, Boyle N, Thao V, Murphy EA, Denzen EM. Perceived Workforce Challenges among Clinical Social Workers in Hematopoietic Cell Transplantation Programs. Biol Blood Marrow Transplant. 2018 May;24(5):1063-1068. doi: 10.1016/j.bbmt.2017.12.793. Epub 2017 Dec 27. PMID 29288820
- [Background] George T, Shah F, Tiwari A, Gutierrez E, Ji J, Kuchel GA, Cohen HJ, Sedrak MS. Resilience in older adults with cancer: A scoping literature review. J Geriatr Oncol. 2023 Jan;14(1):101349. doi: 10.1016/j.jgo.2022.07.009. Epub 2022 Aug 12. PMID 35970715
- [Background] Nakamura ZM, Deal AM, Rosenstein DL, Quillen LJ, Chien SA, Wood WA, Shea TC, Park EM. Cognitive function in patients prior to undergoing allogeneic hematopoietic stem cell transplantation. Support Care Cancer. 2021 Apr;29(4):2007-2014. doi: 10.1007/s00520-020-05697-2. Epub 2020 Aug 23. PMID 32829465
- [Background] Tan JPH, Beilharz JE, Vollmer-Conna U, Cvejic E. Heart rate variability as a marker of healthy ageing. Int J Cardiol. 2019 Jan 15;275:101-103. doi: 10.1016/j.ijcard.2018.08.005. Epub 2018 Aug 3. PMID 30104034
- [Background] Reardon M, Malik M. Changes in heart rate variability with age. Pacing Clin Electrophysiol. 1996 Nov;19(11 Pt 2):1863-6. doi: 10.1111/j.1540-8159.1996.tb03241.x. PMID 8945057
- [Background] Zulfiqar U, Jurivich DA, Gao W, Singer DH. Relation of high heart rate variability to healthy longevity. Am J Cardiol. 2010 Apr 15;105(8):1181-5. doi: 10.1016/j.amjcard.2009.12.022. Epub 2010 Feb 20. PMID 20381674
- [Background] Racioppi A, Dalton T, Ramalingam S, Romero K, Ren Y, Bohannon L, Arellano C, Jonassaint J, Miller H, Barak I, Fish LJ, Choi T, Gasparetto C, Long GD, Lopez RD, Rizzieri DA, Sarantopoulos S, Horwitz ME, Chao NJ, Shah NR, Sung AD. Assessing the Feasibility of a Novel mHealth App in Hematopoietic Stem Cell Transplant Patients. Transplant Cell Ther. 2021 Feb;27(2):181.e1-181.e9. doi: 10.1016/j.jtct.2020.10.017. Epub 2020 Dec 13. PMID 33830035
- [Background] Duking P, Giessing L, Frenkel MO, Koehler K, Holmberg HC, Sperlich B. Wrist-Worn Wearables for Monitoring Heart Rate and Energy Expenditure While Sitting or Performing Light-to-Vigorous Physical Activity: Validation Study. JMIR Mhealth Uhealth. 2020 May 6;8(5):e16716. doi: 10.2196/16716. PMID 32374274
- [Background] Artese AL, Rawat R, Sung AD. The use of commercial wrist-worn technology to track physiological outcomes in behavioral interventions. Curr Opin Clin Nutr Metab Care. 2023 Nov 1;26(6):534-540. doi: 10.1097/MCO.0000000000000970. Epub 2023 Jul 26. PMID 37522804
- [Background] Burton AM, Stock MS. Consistency of novel ultrasound equations for estimating percent intramuscular fat. Clin Physiol Funct Imaging. 2018 Jun 11. doi: 10.1111/cpf.12532. Online ahead of print. PMID 29888525
- [Background] Reimers K, Reimers CD, Wagner S, Paetzke I, Pongratz DE. Skeletal muscle sonography: a correlative study of echogenicity and morphology. J Ultrasound Med. 1993 Feb;12(2):73-7. doi: 10.7863/jum.1993.12.2.73. PMID 8468739
- [Background] Young HJ, Jenkins NT, Zhao Q, Mccully KK. Measurement of intramuscular fat by muscle echo intensity. Muscle Nerve. 2015 Dec;52(6):963-71. doi: 10.1002/mus.24656. Epub 2015 Sep 7. PMID 25787260
- [Background] de Boer AG, Taskila TK, Tamminga SJ, Feuerstein M, Frings-Dresen MH, Verbeek JH. Interventions to enhance return-to-work for cancer patients. Cochrane Database Syst Rev. 2015 Sep 25;2015(9):CD007569. doi: 10.1002/14651858.CD007569.pub3. PMID 26405010
- [Background] Bhatt NS. Prevalence and Determinants of Return to Work as a Patient-Centered Outcome in Survivors of Hematopoietic Cell Transplantation. Curr Hematol Malig Rep. 2022 Dec;17(6):228-242. doi: 10.1007/s11899-022-00678-0. Epub 2022 Oct 4. PMID 36194316
- [Background] Salit RB, Lee SJ, Burns LJ, Shaw BE, Majhail NS, Bhatt NS, Wood WA, Syrjala KL. Return-to-Work Guidelines and Programs for Post-Hematopoietic Cell Transplantation Survivors: An Initial Survey. Biol Blood Marrow Transplant. 2020 Aug;26(8):1520-1526. doi: 10.1016/j.bbmt.2020.04.022. Epub 2020 Apr 29. PMID 32360563
- [Background] van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value Health. 2012 Jul-Aug;15(5):708-15. doi: 10.1016/j.jval.2012.02.008. Epub 2012 May 24. PMID 22867780
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Hahn EA, Beaumont JL, Pilkonis PA, Garcia SF, Magasi S, DeWalt DA, Cella D. The PROMIS satisfaction with social participation measures demonstrated responsiveness in diverse clinical populations. J Clin Epidemiol. 2016 May;73:135-41. doi: 10.1016/j.jclinepi.2015.08.034. Epub 2016 Feb 27. PMID 26931288
- [Background] Khanna D, Maranian P, Rothrock N, Cella D, Gershon R, Khanna PP, Spiegel B, Furst DE, Clements PJ, Bechtel A, Hays RD. Feasibility and construct validity of PROMIS and "legacy" instruments in an academic scleroderma clinic. Value Health. 2012 Jan;15(1):128-34. doi: 10.1016/j.jval.2011.08.006. Epub 2011 Oct 22. PMID 22264980
- [Background] Shensa A, Sidani JE, Escobar-Viera CG, Switzer GE, Primack BA, Choukas-Bradley S. Emotional support from social media and face-to-face relationships: Associations with depression risk among young adults. J Affect Disord. 2020 Jan 1;260:38-44. doi: 10.1016/j.jad.2019.08.092. Epub 2019 Aug 29. PMID 31493637
- [Background] Guerra RS, Fonseca I, Pichel F, Restivo MT, Amaral TF. Usefulness of six diagnostic and screening measures for undernutrition in predicting length of hospital stay: a comparative analysis. J Acad Nutr Diet. 2015 Jun;115(6):927-38. doi: 10.1016/j.jand.2014.11.015. Epub 2015 Jan 27. PMID 25634094
- [Background] Rzepecki P, Barzal J, Sarosiek T, Szczylik C. Biochemical indices for the assessment of nutritional status during hematopoietic stem cell transplantation: are they worth using? A single center experience. Bone Marrow Transplant. 2007 Sep;40(6):567-72. doi: 10.1038/sj.bmt.1705767. Epub 2007 Jul 16. PMID 17637693
- [Background] Espinoza M, Perelli J, Olmos R, Bertin P, Jara V, Ramirez P. Nutritional assessment as predictor of complications after hematopoietic stem cell transplantation. Rev Bras Hematol Hemoter. 2016 Jan-Feb;38(1):7-14. doi: 10.1016/j.bjhh.2015.10.002. Epub 2015 Nov 27. PMID 26969769
- [Background] Urbain P, Birlinger J, Ihorst G, Biesalski HK, Finke J, Bertz H. Body mass index and bioelectrical impedance phase angle as potentially modifiable nutritional markers are independent risk factors for outcome in allogeneic hematopoietic cell transplantation. Ann Hematol. 2013 Jan;92(1):111-9. doi: 10.1007/s00277-012-1573-4. Epub 2012 Sep 12. PMID 22968661
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Clover K, Lambert SD, Oldmeadow C, Britton B, King MT, Mitchell AJ, Carter G. PROMIS depression measures perform similarly to legacy measures relative to a structured diagnostic interview for depression in cancer patients. Qual Life Res. 2018 May;27(5):1357-1367. doi: 10.1007/s11136-018-1803-x. Epub 2018 Feb 8. PMID 29423755
- [Background] Krohe M, Tang DH, Klooster B, Revicki D, Galipeau N, Cella D. Content validity of the National Comprehensive Cancer Network - Functional Assessment of Cancer Therapy - Breast Cancer Symptom Index (NFBSI-16) and Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Short Form with advanced breast cancer patients. Health Qual Life Outcomes. 2019 May 29;17(1):92. doi: 10.1186/s12955-019-1162-5. PMID 31142325
- [Background] Kang JM, Cho YS, Park S, Lee BH, Sohn BK, Choi CH, Choi JS, Jeong HY, Cho SJ, Lee JH, Lee JY. Montreal cognitive assessment reflects cognitive reserve. BMC Geriatr. 2018 Oct 30;18(1):261. doi: 10.1186/s12877-018-0951-8. PMID 30376815
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hill JC, Millan IS. Validation of musculoskeletal ultrasound to assess and quantify muscle glycogen content. A novel approach. Phys Sportsmed. 2014 Sep;42(3):45-52. doi: 10.3810/psm.2014.09.2075. PMID 25295766
- [Background] Baer HR, Thomas SP, Pan Z, Tagawa A, Carollo JJ, Heyn PC. Self-reported physical function is associated with walking speed in adults with cerebral palsy. J Pediatr Rehabil Med. 2019;12(2):181-188. doi: 10.3233/PRM-180585. PMID 31227669
- [Background] Cook KF, Jensen SE, Schalet BD, Beaumont JL, Amtmann D, Czajkowski S, Dewalt DA, Fries JF, Pilkonis PA, Reeve BB, Stone AA, Weinfurt KP, Cella D. PROMIS measures of pain, fatigue, negative affect, physical function, and social function demonstrated clinical validity across a range of chronic conditions. J Clin Epidemiol. 2016 May;73:89-102. doi: 10.1016/j.jclinepi.2015.08.038. Epub 2016 Mar 4. PMID 26952842
- [Background] Moreland JD, Richardson JA, Goldsmith CH, Clase CM. Muscle weakness and falls in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2004 Jul;52(7):1121-9. doi: 10.1111/j.1532-5415.2004.52310.x. PMID 15209650
- [Background] Bieniek J, Wilczynski K, Szewieczek J. Fried frailty phenotype assessment components as applied to geriatric inpatients. Clin Interv Aging. 2016 Apr 22;11:453-9. doi: 10.2147/CIA.S101369. eCollection 2016. PMID 27217729
- [Background] Zhang Q, Li YX, Li XL, Yin Y, Li RL, Qiao X, Li W, Ma HF, Ma WH, Han YF, Zeng GQ, Wang QY, Kang J, Hou G. A comparative study of the five-repetition sit-to-stand test and the 30-second sit-to-stand test to assess exercise tolerance in COPD patients. Int J Chron Obstruct Pulmon Dis. 2018 Sep 10;13:2833-2839. doi: 10.2147/COPD.S173509. eCollection 2018. PMID 30237707
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Lauretani F, Ticinesi A, Gionti L, Prati B, Nouvenne A, Tana C, Meschi T, Maggio M. Short-Physical Performance Battery (SPPB) score is associated with falls in older outpatients. Aging Clin Exp Res. 2019 Oct;31(10):1435-1442. doi: 10.1007/s40520-018-1082-y. Epub 2018 Dec 4. PMID 30515724
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Adachi H. Cardiopulmonary Exercise Test. Int Heart J. 2017 Oct 21;58(5):654-665. doi: 10.1536/ihj.17-264. Epub 2017 Sep 30. PMID 28966333
- [Background] Vandekerckhove K, De Waele K, Minne A, Coomans I, De Groote K, Panzer J, Dhooge C, Bordon V, De Wolf D, Boone J. Evaluation of cardiopulmonary exercise testing, heart function, and quality of life in children after allogenic hematopoietic stem cell transplantation. Pediatr Blood Cancer. 2019 Jan;66(1):e27499. doi: 10.1002/pbc.27499. Epub 2018 Oct 14. PMID 30318730
- [Background] Mishra A, Pidala J, Thapa R, Betts BC, Fernandez H, Locke FL, Nishihori T, Perez L, Wang X, Anasetti C, Jim H. Objective and subjective physical function in allogeneic hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2021 Dec;56(12):2897-2903. doi: 10.1038/s41409-021-01428-1. Epub 2021 Aug 11. PMID 34381169
- [Background] Penna GB, da Silva TC, Aparecida Paz A, Ziegler B. Functional capacity, pulmonary function, and quality of life in hematopoietic stem cell transplantation survivors. Support Care Cancer. 2021 Jul;29(7):4015-4021. doi: 10.1007/s00520-020-05947-3. Epub 2021 Jan 4. PMID 33394196
- [Background] Enright PL. The six-minute walk test. Respir Care. 2003 Aug;48(8):783-5. PMID 12890299
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Schoenmakers PPJM, Hettinga FJ, Reed KE. The Moderating Role of Recovery Durations in High-Intensity Interval-Training Protocols. Int J Sports Physiol Perform. 2019 Jul 1;14(6):859-867. doi: 10.1123/ijspp.2018-0876. PMID 31146621
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Wood WA, Deal AM, Reeve BB, Abernethy AP, Basch E, Mitchell SA, Shatten C, Hie Kim Y, Whitley J, Serody JS, Shea T, Battaglini C. Cardiopulmonary fitness in patients undergoing hematopoietic SCT: a pilot study. Bone Marrow Transplant. 2013 Oct;48(10):1342-9. doi: 10.1038/bmt.2013.58. Epub 2013 Apr 15. PMID 23584437
- [Background] Coleman EA, Coon SK, Kennedy RL, Lockhart KD, Stewart CB, Anaissie EJ, Barlogie B. Effects of exercise in combination with epoetin alfa during high-dose chemotherapy and autologous peripheral blood stem cell transplantation for multiple myeloma. Oncol Nurs Forum. 2008 May;35(3):E53-61. doi: 10.1188/08.ONF.E53-E61. PMID 18467280
- [Background] Wood WA, Phillips B, Smith-Ryan AE, Wilson D, Deal AM, Bailey C, Meeneghan M, Reeve BB, Basch EM, Bennett AV, Shea TC, Battaglini CL. Personalized home-based interval exercise training may improve cardiorespiratory fitness in cancer patients preparing to undergo hematopoietic cell transplantation. Bone Marrow Transplant. 2016 Jul;51(7):967-72. doi: 10.1038/bmt.2016.73. Epub 2016 Mar 21. PMID 26999467
- [Background] Wood WA, Weaver M, Smith-Ryan AE, Hanson ED, Shea TC, Battaglini CL. Lessons learned from a pilot randomized clinical trial of home-based exercise prescription before allogeneic hematopoietic cell transplantation. Support Care Cancer. 2020 Nov;28(11):5291-5298. doi: 10.1007/s00520-020-05369-1. Epub 2020 Feb 28. PMID 32112353
- [Background] Santa Mina D, Dolan LB, Lipton JH, Au D, Camacho Perez E, Franzese A, Alibhai SMH, Jones JM, Chang E. Exercise before, during, and after Hospitalization for Allogeneic Hematological Stem Cell Transplant: A Feasibility Randomized Controlled Trial. J Clin Med. 2020 Jun 14;9(6):1854. doi: 10.3390/jcm9061854. PMID 32545872
- [Background] Persoon S, Kersten MJ, van der Weiden K, Buffart LM, Nollet F, Brug J, Chinapaw MJ. Effects of exercise in patients treated with stem cell transplantation for a hematologic malignancy: a systematic review and meta-analysis. Cancer Treat Rev. 2013 Oct;39(6):682-90. doi: 10.1016/j.ctrv.2013.01.001. Epub 2013 Feb 26. PMID 23485478
- [Background] Canestraro A, Nakhle A, Stack M, Strong K, Wright A, Beauchamp M, Berg K, Brooks D. Oncology Rehabilitation Provision and Practice Patterns across Canada. Physiother Can. 2013 Winter;65(1):94-102. doi: 10.3138/ptc.2011-53. PMID 24381389
- [Background] Parker NH, Arlinghaus KR, Johnston CA. Integrating Physical Activity Into Clinical Cancer Care. Am J Lifestyle Med. 2018 Mar 5;12(3):220-223. doi: 10.1177/1559827618759478. eCollection 2018 May-Jun. PMID 30283253
- [Background] Falkenburg JHF, Jedema I. Graft versus tumor effects and why people relapse. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):693-698. doi: 10.1182/asheducation-2017.1.693. PMID 29222323
- [Background] Sweeney C, Vyas P. The Graft-Versus-Leukemia Effect in AML. Front Oncol. 2019 Nov 19;9:1217. doi: 10.3389/fonc.2019.01217. eCollection 2019. PMID 31803612
- [Background] Cieri N, Mastaglio S, Oliveira G, Casucci M, Bondanza A, Bonini C. Adoptive immunotherapy with genetically modified lymphocytes in allogeneic stem cell transplantation. Immunol Rev. 2014 Jan;257(1):165-80. doi: 10.1111/imr.12130. PMID 24329796
- [Background] Soiffer R. Immune modulation and chronic graft-versus-host disease. Bone Marrow Transplant. 2008 Aug;42 Suppl 1:S66-S69. doi: 10.1038/bmt.2008.119. PMID 18724307
- [Background] Robinson E, Durrer C, Simtchouk S, Jung ME, Bourne JE, Voth E, Little JP. Short-term high-intensity interval and moderate-intensity continuous training reduce leukocyte TLR4 in inactive adults at elevated risk of type 2 diabetes. J Appl Physiol (1985). 2015 Sep 1;119(5):508-16. doi: 10.1152/japplphysiol.00334.2015. Epub 2015 Jul 2. PMID 26139217
- [Background] Bartlett DB, Duggal NA. Moderate physical activity associated with a higher naive/memory T-cell ratio in healthy old individuals: potential role of IL15. Age Ageing. 2020 Apr 27;49(3):368-373. doi: 10.1093/ageing/afaa035. PMID 32221610
- [Background] Duggal NA, Pollock RD, Lazarus NR, Harridge S, Lord JM. Major features of immunesenescence, including reduced thymic output, are ameliorated by high levels of physical activity in adulthood. Aging Cell. 2018 Apr;17(2):e12750. doi: 10.1111/acel.12750. Epub 2018 Mar 8. PMID 29517845
- [Background] Duggal NA, Niemiro G, Harridge SDR, Simpson RJ, Lord JM. Can physical activity ameliorate immunosenescence and thereby reduce age-related multi-morbidity? Nat Rev Immunol. 2019 Sep;19(9):563-572. doi: 10.1038/s41577-019-0177-9. PMID 31175337
- [Background] Biazus-Sehn LF, Schuch FB, Firth J, Stigger FS. Effects of physical exercise on cognitive function of older adults with mild cognitive impairment: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2020 Jul-Aug;89:104048. doi: 10.1016/j.archger.2020.104048. Epub 2020 May 12. PMID 32460123
- [Background] Ehlers DK, Aguinaga S, Cosman J, Severson J, Kramer AF, McAuley E. The effects of physical activity and fatigue on cognitive performance in breast cancer survivors. Breast Cancer Res Treat. 2017 Oct;165(3):699-707. doi: 10.1007/s10549-017-4363-9. Epub 2017 Jul 4. PMID 28677009
- [Background] Liu PZ, Nusslock R. Exercise-Mediated Neurogenesis in the Hippocampus via BDNF. Front Neurosci. 2018 Feb 7;12:52. doi: 10.3389/fnins.2018.00052. eCollection 2018. PMID 29467613
- [Background] Morales-Rodriguez E, Perez-Bilbao T, San Juan AF, Calvo JL. Effects of Exercise Programs on Physical Factors and Safety in Adult Patients with Cancer and Haematopoietic Stem Cell Transplantation: A Systematic Review. Int J Environ Res Public Health. 2022 Jan 24;19(3):1288. doi: 10.3390/ijerph19031288. PMID 35162312
- [Background] Fiuza-Luces C, Simpson RJ, Ramirez M, Lucia A, Berger NA. Physical function and quality of life in patients with chronic GvHD: a summary of preclinical and clinical studies and a call for exercise intervention trials in patients. Bone Marrow Transplant. 2016 Jan;51(1):13-26. doi: 10.1038/bmt.2015.195. Epub 2015 Sep 14. PMID 26367233
- [Background] Morales Rodriguez E, Lorenzo Calvo J, Granado-Peinado M, Perez-Bilbao T, San Juan AF. Effects of Exercise Programs on Psychoemotional and Quality-of-Life Factors in Adult Patients with Cancer and Hematopoietic Stem Cell Transplantation or Bone Marrow Transplantation: A Systematic Review. Int J Environ Res Public Health. 2022 Nov 29;19(23):15896. doi: 10.3390/ijerph192315896. PMID 36497971
- [Background] Leach HJ, Danyluk JM, Nishimura KC, Culos-Reed SN. Benefits of 24 versus 12 weeks of exercise and wellness programming for women undergoing treatment for breast cancer. Support Care Cancer. 2016 Nov;24(11):4597-606. doi: 10.1007/s00520-016-3302-3. Epub 2016 Jun 16. PMID 27312845
- [Background] Koevoets EW, Schagen SB, de Ruiter MB, Geerlings MI, Witlox L, van der Wall E, Stuiver MM, Sonke GS, Velthuis MJ, Jobsen JJ, Menke-Pluijmers MBE, Goker E, van der Pol CC, Bos MEMM, Tick LW, van Holsteijn NA, van der Palen J, May AM, Monninkhof EM; PAM study group. Effect of physical exercise on cognitive function after chemotherapy in patients with breast cancer: a randomized controlled trial (PAM study). Breast Cancer Res. 2022 May 26;24(1):36. doi: 10.1186/s13058-022-01530-2. PMID 35619188
- [Background] Abo S, Denehy L, Ritchie D, Lin KY, Edbrooke L, McDonald C, Granger CL. People With Hematological Malignancies Treated With Bone Marrow Transplantation Have Improved Function, Quality of Life, and Fatigue Following Exercise Intervention: A Systematic Review and Meta-Analysis. Phys Ther. 2021 Aug 1;101(8):pzab130. doi: 10.1093/ptj/pzab130. PMID 33989413
- [Background] van Haren IE, Timmerman H, Potting CM, Blijlevens NM, Staal JB, Nijhuis-van der Sanden MW. Physical exercise for patients undergoing hematopoietic stem cell transplantation: systematic review and meta-analyses of randomized controlled trials. Phys Ther. 2013 Apr;93(4):514-28. doi: 10.2522/ptj.20120181. Epub 2012 Dec 6. PMID 23224217
- [Background] Singh B, Hayes SC, Spence RR, Steele ML, Millet GY, Gergele L. Exercise and colorectal cancer: a systematic review and meta-analysis of exercise safety, feasibility and effectiveness. Int J Behav Nutr Phys Act. 2020 Sep 24;17(1):122. doi: 10.1186/s12966-020-01021-7. PMID 32972439
- [Background] Myers JS, Erickson KI, Sereika SM, Bender CM. Exercise as an Intervention to Mitigate Decreased Cognitive Function From Cancer and Cancer Treatment: An Integrative Review. Cancer Nurs. 2018 Jul/Aug;41(4):327-343. doi: 10.1097/NCC.0000000000000549. PMID 29194066
- [Background] Misiag W, Piszczyk A, Szymanska-Chabowska A, Chabowski M. Physical Activity and Cancer Care-A Review. Cancers (Basel). 2022 Aug 27;14(17):4154. doi: 10.3390/cancers14174154. PMID 36077690
- [Background] Sitlinger A, Brander DM, Bartlett DB. Impact of exercise on the immune system and outcomes in hematologic malignancies. Blood Adv. 2020 Apr 28;4(8):1801-1811. doi: 10.1182/bloodadvances.2019001317. PMID 32343800
- [Background] Knips L, Bergenthal N, Streckmann F, Monsef I, Elter T, Skoetz N. Aerobic physical exercise for adult patients with haematological malignancies. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD009075. doi: 10.1002/14651858.CD009075.pub3. PMID 30702150
- [Background] Young J, Angevaren M, Rusted J, Tabet N. Aerobic exercise to improve cognitive function in older people without known cognitive impairment. Cochrane Database Syst Rev. 2015 Apr 22;2015(4):CD005381. doi: 10.1002/14651858.CD005381.pub4. PMID 25900537
- [Background] Argent R, Daly A, Caulfield B. Patient Involvement With Home-Based Exercise Programs: Can Connected Health Interventions Influence Adherence? JMIR Mhealth Uhealth. 2018 Mar 1;6(3):e47. doi: 10.2196/mhealth.8518. PMID 29496655
- [Background] Paterson DH, Cunningham DA, Koval JJ, St Croix CM. Aerobic fitness in a population of independently living men and women aged 55-86 years. Med Sci Sports Exerc. 1999 Dec;31(12):1813-20. doi: 10.1097/00005768-199912000-00018. PMID 10613433
- [Background] Sasso JP, Eves ND, Christensen JF, Koelwyn GJ, Scott J, Jones LW. A framework for prescription in exercise-oncology research. J Cachexia Sarcopenia Muscle. 2015 Jun;6(2):115-24. doi: 10.1002/jcsm.12042. Epub 2015 May 11. PMID 26136187
- [Background] Wong JN, McAuley E, Trinh L. Physical activity programming and counseling preferences among cancer survivors: a systematic review. Int J Behav Nutr Phys Act. 2018 Jun 7;15(1):48. doi: 10.1186/s12966-018-0680-6. PMID 29879993
- [Background] Shepherd SO, Wilson OJ, Taylor AS, Thogersen-Ntoumani C, Adlan AM, Wagenmakers AJ, Shaw CS. Low-Volume High-Intensity Interval Training in a Gym Setting Improves Cardio-Metabolic and Psychological Health. PLoS One. 2015 Sep 24;10(9):e0139056. doi: 10.1371/journal.pone.0139056. eCollection 2015. PMID 26402859
- [Background] Campbell WW, Kraus WE, Powell KE, Haskell WL, Janz KF, Jakicic JM, Troiano RP, Sprow K, Torres A, Piercy KL, Bartlett DB; 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. High-Intensity Interval Training for Cardiometabolic Disease Prevention. Med Sci Sports Exerc. 2019 Jun;51(6):1220-1226. doi: 10.1249/MSS.0000000000001934. PMID 31095079
- [Background] Bartlett DB, Willis LH, Slentz CA, Hoselton A, Kelly L, Huebner JL, Kraus VB, Moss J, Muehlbauer MJ, Spielmann G, Kraus WE, Lord JM, Huffman KM. Ten weeks of high-intensity interval walk training is associated with reduced disease activity and improved innate immune function in older adults with rheumatoid arthritis: a pilot study. Arthritis Res Ther. 2018 Jun 14;20(1):127. doi: 10.1186/s13075-018-1624-x. PMID 29898765
- [Background] Bartlett DB, Slentz CA, Willis LH, Hoselton A, Huebner JL, Kraus VB, Moss J, Muehlbauer MJ, Spielmann G, Muoio DM, Koves TR, Wu H, Huffman KM, Lord JM, Kraus WE. Rejuvenation of Neutrophil Functions in Association With Reduced Diabetes Risk Following Ten Weeks of Low-Volume High Intensity Interval Walking in Older Adults With Prediabetes - A Pilot Study. Front Immunol. 2020 May 5;11:729. doi: 10.3389/fimmu.2020.00729. eCollection 2020. PMID 32431698
- [Background] Bartlett DB, Shepherd SO, Wilson OJ, Adlan AM, Wagenmakers AJM, Shaw CS, Lord JM. Neutrophil and Monocyte Bactericidal Responses to 10 Weeks of Low-Volume High-Intensity Interval or Moderate-Intensity Continuous Training in Sedentary Adults. Oxid Med Cell Longev. 2017;2017:8148742. doi: 10.1155/2017/8148742. Epub 2017 Jun 1. PMID 28656073
- [Background] Artese AL, Winthrop HM, Bohannon L, Lew MV, Johnson E, MacDonald G, Ren Y, Pastva AM, Hall KS, Wischmeyer PE, Macleod D, Molinger J, Barth S, Jung SH, Cohen HJ, Bartlett DB, Sung AD. A pilot study to assess the feasibility of a remotely monitored high-intensity interval training program prior to allogeneic hematopoietic stem cell transplantation. PLoS One. 2023 Nov 30;18(11):e0293171. doi: 10.1371/journal.pone.0293171. eCollection 2023. PMID 38032994
- [Background] Wingard JR, Wood WA, Martens M, Le-Rademacher J, Logan B, Knight JM, Jacobsen PB, Jim H, Majhail NS, Syrjala K, Rizzo JD, Lee SJ. Pretransplantation Exercise and Hematopoietic Cell Transplantation Survival: A Secondary Analysis of Blood and Marrow Transplant Clinical Trials Network (BMT CTN 0902). Biol Blood Marrow Transplant. 2017 Jan;23(1):161-164. doi: 10.1016/j.bbmt.2016.10.007. Epub 2016 Oct 11. PMID 27742574
- [Background] Wiskemann J, Kleindienst N, Kuehl R, Dreger P, Schwerdtfeger R, Bohus M. Effects of physical exercise on survival after allogeneic stem cell transplantation. Int J Cancer. 2015 Dec 1;137(11):2749-56. doi: 10.1002/ijc.29633. Epub 2015 Jun 19. PMID 26061092
- [Background] Min GJ, Cho BS, Kwag D, Park SS, Park S, Yoon JH, Lee SE, Eom KS, Kim YJ, Lee S, Min CK, Cho SG, Lee JW, Kim HJ. Dynamic changes in physical function during intensive chemotherapy affect transplant outcomes in older adults with AML. Front Oncol. 2023 Nov 7;13:1281782. doi: 10.3389/fonc.2023.1281782. eCollection 2023. PMID 38023260
- [Background] De Lisio M, Parise G. Exercise and hematopoietic stem and progenitor cells: protection, quantity, and function. Exerc Sport Sci Rev. 2013 Apr;41(2):116-22. doi: 10.1097/JES.0b013e3182877deb. PMID 23364348
- [Background] De Lisio M, Baker JM, Parise G. Exercise promotes bone marrow cell survival and recipient reconstitution post-bone marrow transplantation, which is associated with increased survival. Exp Hematol. 2013 Feb;41(2):143-54. doi: 10.1016/j.exphem.2012.10.003. Epub 2012 Oct 11. PMID 23063724
- [Background] El-Jawahri A, LeBlanc T, VanDusen H, Traeger L, Greer JA, Pirl WF, Jackson VA, Telles J, Rhodes A, Spitzer TR, McAfee S, Chen YA, Lee SS, Temel JS. Effect of Inpatient Palliative Care on Quality of Life 2 Weeks After Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2016 Nov 22;316(20):2094-2103. doi: 10.1001/jama.2016.16786. PMID 27893130
- [Background] El-Jawahri A, Traeger L, Greer JA, VanDusen H, Fishman SR, LeBlanc TW, Pirl WF, Jackson VA, Telles J, Rhodes A, Li Z, Spitzer TR, McAfee S, Chen YA, Temel JS. Effect of Inpatient Palliative Care During Hematopoietic Stem-Cell Transplant on Psychological Distress 6 Months After Transplant: Results of a Randomized Clinical Trial. J Clin Oncol. 2017 Nov 10;35(32):3714-3721. doi: 10.1200/JCO.2017.73.2800. Epub 2017 Sep 19. PMID 28926288
- [Background] Andorsky DJ, Loberiza FR, Lee SJ. Pre-transplantation physical and mental functioning is strongly associated with self-reported recovery from stem cell transplantation. Bone Marrow Transplant. 2006 May;37(9):889-95. doi: 10.1038/sj.bmt.1705347. PMID 16532014
- [Background] Bevans M, El-Jawahri A, Tierney DK, Wiener L, Wood WA, Hoodin F, Kent EE, Jacobsen PB, Lee SJ, Hsieh MM, Denzen EM, Syrjala KL. National Institutes of Health Hematopoietic Cell Transplantation Late Effects Initiative: The Patient-Centered Outcomes Working Group Report. Biol Blood Marrow Transplant. 2017 Apr;23(4):538-551. doi: 10.1016/j.bbmt.2016.09.011. Epub 2016 Sep 19. PMID 27660168
- [Background] Jones LW, Devlin SM, Maloy MA, Wood WA, Tuohy S, Espiritu N, Aquino J, Kendig T, Michalski MG, Gyurkocza B, Schaffer WL, Ali B, Giralt S, Jakubowski AA. Prognostic Importance of Pretransplant Functional Capacity After Allogeneic Hematopoietic Cell Transplantation. Oncologist. 2015 Nov;20(11):1290-7. doi: 10.1634/theoncologist.2015-0200. Epub 2015 Oct 7. PMID 26446235
- [Background] Wood WA, Le-Rademacher J, Syrjala KL, Jim H, Jacobsen PB, Knight JM, Abidi MH, Wingard JR, Majhail NS, Geller NL, Rizzo JD, Fei M, Wu J, Horowitz MM, Lee SJ. Patient-reported physical functioning predicts the success of hematopoietic cell transplantation (BMT CTN 0902). Cancer. 2016 Jan 1;122(1):91-8. doi: 10.1002/cncr.29717. Epub 2015 Oct 6. PMID 26439325
- [Background] Steinberg A, Asher A, Bailey C, Fu JB. The role of physical rehabilitation in stem cell transplantation patients. Support Care Cancer. 2015 Aug;23(8):2447-60. doi: 10.1007/s00520-015-2744-3. Epub 2015 May 14. PMID 25971213
- [Background] Dimeo FC, Stieglitz RD, Novelli-Fischer U, Fetscher S, Keul J. Effects of physical activity on the fatigue and psychologic status of cancer patients during chemotherapy. Cancer. 1999 May 15;85(10):2273-7. PMID 10326708
- [Background] Pamukcuoglu M, Bhatia S, Weisdorf DJ, DeFor TE, Ustun C, Nayar M, Holtan SG, Jurdi NE, Thyagarajan B, Brunstein CG, Bachanova V, Warlick ED, Severseike B, Te HS, Lund T, Arora M. Hematopoietic Cell Transplant-Related Toxicities and Mortality in Frail Recipients. Biol Blood Marrow Transplant. 2019 Dec;25(12):2454-2460. doi: 10.1016/j.bbmt.2019.07.030. Epub 2019 Aug 5. PMID 31394273
- [Background] Hacker ED. Physical Activity and Exercise after Hematopoietic Cell Transplantation: Just Keep on Moving. Asia Pac J Oncol Nurs. 2019 Jan-Mar;6(1):1-3. doi: 10.4103/apjon.apjon_64_18. No abstract available. PMID 30599007
- [Background] Penack O, Peczynski C, Mohty M, Yakoub-Agha I, Styczynski J, Montoto S, Duarte RF, Kroger N, Schoemans H, Koenecke C, Peric Z, Basak GW. How much has allogeneic stem cell transplant-related mortality improved since the 1980s? A retrospective analysis from the EBMT. Blood Adv. 2020 Dec 22;4(24):6283-6290. doi: 10.1182/bloodadvances.2020003418. PMID 33351121
- [Background] Gooley TA, Chien JW, Pergam SA, Hingorani S, Sorror ML, Boeckh M, Martin PJ, Sandmaier BM, Marr KA, Appelbaum FR, Storb R, McDonald GB. Reduced mortality after allogeneic hematopoietic-cell transplantation. N Engl J Med. 2010 Nov 25;363(22):2091-101. doi: 10.1056/NEJMoa1004383. PMID 21105791
- [Background] Horan JT, Logan BR, Agovi-Johnson MA, Lazarus HM, Bacigalupo AA, Ballen KK, Bredeson CN, Carabasi MH, Gupta V, Hale GA, Khoury HJ, Juckett MB, Litzow MR, Martino R, McCarthy PL, Smith FO, Rizzo JD, Pasquini MC. Reducing the risk for transplantation-related mortality after allogeneic hematopoietic cell transplantation: how much progress has been made? J Clin Oncol. 2011 Mar 1;29(7):805-13. doi: 10.1200/JCO.2010.32.5001. Epub 2011 Jan 10. PMID 21220593
- [Background] Robin M, Porcher R, Ades L, Boissel N, Raffoux E, Xhaard A, Larghero J, Gardin C, Himberlin C, Delmer A, Fenaux P, Dombret H, Socie G, Peffault de Latour R. Matched unrelated or matched sibling donors result in comparable outcomes after non-myeloablative HSCT in patients with AML or MDS. Bone Marrow Transplant. 2013 Oct;48(10):1296-301. doi: 10.1038/bmt.2013.50. Epub 2013 Apr 15. PMID 23584440
- [Background] 3. Bolon YT AR, Allbee-Johnson M, Estrada-Merly N, Lee SJ. . Current use and outcome of hematopoietic stem cell transplantation: CIBMTR summary slides,2022
- [Background] Perales MA, Bonafede M, Cai Q, Garfin PM, McMorrow D, Josephson NC, Richhariya A. Real-World Economic Burden Associated with Transplantation-Related Complications. Biol Blood Marrow Transplant. 2017 Oct;23(10):1788-1794. doi: 10.1016/j.bbmt.2017.06.017. Epub 2017 Jul 5. PMID 28688917
- [Background] D'Souza A, Fretham C, Lee SJ, Arora M, Brunner J, Chhabra S, Devine S, Eapen M, Hamadani M, Hari P, Pasquini MC, Perez W, Phelan RA, Riches ML, Rizzo JD, Saber W, Shaw BE, Spellman SR, Steinert P, Weisdorf DJ, Horowitz MM. Current Use of and Trends in Hematopoietic Cell Transplantation in the United States. Biol Blood Marrow Transplant. 2020 Aug;26(8):e177-e182. doi: 10.1016/j.bbmt.2020.04.013. Epub 2020 May 11. PMID 32438042